CLINICAL TRIAL: NCT05633433
Title: A Phase II/III Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Individuals Infected With SARS-CoV-2
Brief Title: Evaluate the Efficacy and Safety of Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Covid-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry); Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FNC-Covid304
Record Dates: First submitted 2022-11-30; First posted 2022-12-01 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — azvudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- cohort A （Phase II） (Experimental): Azvudine 5 mg, QD PO, D1-D7
  Interventions: Drug: Azvudine
- cohort B （Phase II） (Experimental): Azvudine 3 mg + placebo 2 mg, QD PO, D1-D7
  Interventions: Drug: Azvudine; Drug: Placebo
- cohort C （Phase II） (Placebo Comparator): placebo 5 mg, QD PO, D1-D7
  Interventions: Drug: Placebo
- Arm 1 (Phase III) (Experimental): Azvudine, dose to be determined according to phase II, QD PO, D1-D7
  Interventions: Drug: Azvudine
- Arm 2 (Phase III) (Placebo Comparator): Placebo, dose to be the same as Arm1, QD PO, D1-D7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azvudine — Azvudine is a novel nucleoside reverse transcriptase inhibitor.
  Other Names: FNC
  Arms: Arm 1 (Phase III); cohort A （Phase II）; cohort B （Phase II）
Drug: Placebo — Placebo
  Arms: Arm 2 (Phase III); cohort B （Phase II）; cohort C （Phase II）

SUMMARY:
A Phase II/III Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Individuals Infected with SARS-CoV-2

DETAILED DESCRIPTION:
The study has two parts:

Part 1 is a multicentre, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of Azvudine versus placebo in preventing SARS-CoV-2 infection in household contacts with SARS-CoV-2 infection individuals. The population of part 1 will consist of approximately 450 adults with household contact exposure to individuals with a confirmed SARS-CoV-2 infection.A phase III study will be further conducted if any of the treatment groups reduce SARS-CoV-2 infection rate (Relative risk reduction) > 50% compared with the placebo group.

Part 2 is a multicentre, randomized, double-blind, placebo-controlled phase III clinical study. The subject sample size will be calculated based on the results of the Phase II trial.

Phase II and phase III studies have the same objectives and primary/secondary end points. The primary endpoint is the proportion of subjects with positive SARS-CoV-2 RT-PCR assay in 7 days. Nasopharyngeal swabs will be collected at D2, D4, D7, D10, and D14 by RT-PCR to confirm SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old at the signing of informed consent.
2. Household contacts of individual with symptomatic COVID-19. Symptomatic COVID-19 cases (index case) to be identified as those symptomatic and recently tested (rapid antigen test or RT-PCR) positive for SARS-CoV-2 and must fulfill the following criteria 1) collection of the first positive SARS-CoV-2 test sample less than 48 hours before randomization, 2) have at least one symptom attributable to COVID-19.
3. RT-PCR test negative (with nasopharyngeal [NP] swab samples) OR rapid antigen test negative at the time of screening and without any suspicious COVID-19 symptoms within 2 weeks before randomization.
4. Subject expects to be living in the same household with the symptomatic COVID-19 cases during the whole study period.
5. Willing and able to comply with study visits and study-related procedures/assessments.
6. Provide informed consent signed by study subject or legally acceptable representative.

Exclusion Criteria:

1. Subject with a history of SARS-CoV-2 vaccinations within 6 months before randomization.
2. Subject with a history of SARS-CoV-2 infection within 6 months before randomization.
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3×Upper Limit of Normal (ULN) ,or total bilirubin (TBIL) >2×ULN.
4. Creatinine clearance (Ccr, calculated by Cockcroft-Gault equation)<60 ml/min or Creatinine >1.2×ULN.
5. With any serious infection requiring systemic anti-infective therapy within 14 days before randomization.
6. Allergic to the investigational agent or any components of the formulation.
7. Pregnant or breast-feeding women.
8. Previous administration of any antiretroviral drugs (e.g., antiretroviral drugs for HIV, HBV, or HCV) within 7 days before randomization.
9. Women of childbearing potential who are unwilling to practice highly effective contraception during the study, and for at least 6 months after the study; Sexually active men who are unwilling to use medically acceptable birth control during the study period.
10. Have other conditions not suitable for inclusion as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Incidence of SARS-CoV-2 infection in 7 days | Day 2 to Day 7
  The incidence of SARS-CoV-2 infection (RT-PCR positive) up to 7 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.

SECONDARY OUTCOMES:
Incidence of asymptomatic SARS-CoV-2 infection in 7 days | Day 2 to Day 7
  The incidence of asymptomatic SARS-CoV-2 infection (RT-PCR positive) up to 7 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of symptomatic SARS-CoV-2 infection in 7 days | Day 2 to Day 7
  The incidence of symptomatic SARS-CoV-2 infection (RT-PCR positive) up to 7 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of SARS-CoV-2 infection in 14 days | Day 2 to Day 14
  The incidence of SARS-CoV-2 infection (RT-PCR positive) up to 14 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of asymptomatic SARS-CoV-2 infection in 14 days | Day 2 to Day 14
  The incidence of asymptomatic SARS-CoV-2 infection (RT-PCR positive) up to 14 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of symptomatic SARS-CoV-2 infection in 14 days | Day 2 to Day 14
  The incidence of SARS-CoV-2 infection (RT-PCR positive) up to 14 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of severe COVID-19 | Day 1 to Day 28
  To describe the incidence of severe COVID-19 up to 28 days after administration of Azvudine for prevention of SARS-CoV-2 infection.
Incidence of all-cause mortality | Day 1 to Day 28
  To describe the incidence of all-cause mortality during the 28 days after administration of Azvudine for prevention of SAR-CoV-2 infection.
Time to SARS-CoV-2 infection | Day 1 to Day 28
  The time to SARS-CoV-2 infection after the the first dose of Azvudine will be evaluated in the RT-PCR positive participants.
Duration of symptoms | Day 1 to Day 28
  Duration of symptoms in participants with COVID-19.
Adverse events | Day 1 to Day 28
  Number of participants with adverse events after administration of Azvudine will be evaluated.
Maximum serum concentration (Cmax) | Day 1 to Day 28
  The Cmax of Azvudine after administration in participants will be evaluated.
Time to reach maximum serum concentration (Tmax) | Day 1 to Day 28
  The Tmax of Azvudine after administration in participants will be evaluated.
Terminal half-life (T1/2) | Day 1 to Day 28
  The T1/2 of Azvudine after administration in participants will be evaluated.
Apparent total clearance (CL/F) | Day 1 to Day 28
  The CL/F of Azvudine after administration in participants will be evaluated.
Apparent volume of distribution based on terminal phase (Vz/F) | Day 1 to Day 28
  The Vz/F of Azvudine after administration in participants will be evaluated.
Area under the concentration-time curve from time 0 to the last concentration-measurable time point (AUC0-t) | Day 1 to Day 28
  The AUC0-t of Azvudine after administration in participants will be evaluated.
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) | Day 1 to Day 28
  The AUC0-∞ of Azvudine after administration in participants will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard S. Garcia, M.D., Principal Investigator — Cebu Doctor's University Hospital
Locations (10):
- Malaysia (7):
  - University of Malaya Medical Centre, Kuala Lumpur
  - International Islamic University Malaysia, Kuantan
  - ALPS Medical Center, Shah Alam
  - Klinik Kesihatan Cheras, Shah Alam
  - Klinik Kesihatan Greentown, Shah Alam
  - Klinik Kesihatan Kuala Kedah, Shah Alam
  - Klinik Kesihatan Mahmoodiah, Shah Alam
- Philippines (3):
  - Cebu Doctors' University Hospitol, Cebu City
  - Perpetual Succour Hospital, Cebu City
  - University of the East Ramon Magsaysay Memorial Medical Center, Quezon City

IPD SHARING:
Plan to Share IPD: No